CLINICAL TRIAL: NCT06127654
Title: VITaL: A Randomised Controlled Trial Investigating Ventilation Imaging to Improve the Quality of Life for Patients With Lung Cancer Treated With Radiation Therapy
Brief Title: Ventilation Imaging to Improve the Quality of Life for Patients With Lung Cancer Treated With Radiation Therapy
Acronym: VITaL
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Liverpool Hospital (Unknown); Royal North Shore Hospital (Other); The Alfred (Other); Peter MacCallum Cancer Centre, Australia (Other); Fundacion GenesisCare (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IX-2022-CT-VITAL
Record Dates: First submitted 2023-10-30; First posted 2023-11-13 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer
Keywords: Pneumonitis; Quality of Life; Curative treatment; Cancer; Healthy lung sparing
MeSH Terms: conditions — Lung Neoplasms; Pneumonia; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Lung sparing treatment plan
  Interventions: Device: Healthy lung sparing treatment plan
- Control (No Intervention): Standard treatment plan

INTERVENTIONS:
Device: Healthy lung sparing treatment plan — CT Ventilation imaging will be used to create a healthy lung sparing treatment plan for patients who will receive radiation therapy treatment for their lung cancer.
  Arms: Intervention

SUMMARY:
This research project is testing a new treatment planning method for patients with lung cancer who will be treated with radiation therapy. This new method is called Computed Tomography (CT) ventilation imaging. It aims to help protect the healthiest parts of patient's lungs from being injured by the radiation therapy. The investigators will determine whether healthy lung sparing can improve the quality of life in these patients.

DETAILED DESCRIPTION:
The planning and delivery of Radiation Therapy (RT) is a balance between delivering a curative dose to the tumour while sparing healthy organs, such as the lungs, from collateral damage such as pneumonitis. To minimise radiation-induced lung injury, our team has invented and pioneered ventilation imaging based on Computed Tomography (CT). This Australian-invented medical device, now an international field of research, uses CT scans routinely acquired for planning RT to compute a CT ventilation map showing high functioning and low functioning lung regions. This image is used as the basis for directing radiation away from the healthy, high functioning regions towards the low functioning regions, thereby aiming to reduce toxicity and improve the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria

1. Aged 18 years or older.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
3. Histologically proven non-small cell lung cancer.
4. Stage 3 as determined using the IASLC (International Association for the Study of Lung Cancer) 8th edition lung cancer staging guidelines.
5. To be treated with curative intent external beam radiotherapy (60 Gy in 30 treatments or 55 Gy in 20 treatments) +/- concurrent chemotherapy and adjuvant PD1/PD-L1 inhibitors.
6. Whole body Positron Emission Tomography (PET) scan within 8 weeks of registration.
7. Pulmonary function tests within 8 weeks of registration.
8. Willingness to give written informed consent.
9. Willingness to comply with the study procedures and visit requirements.
10. Available for follow up for a minimum of 12 months and up to 3 years.

Post-inclusion criteria includes the results of a Quality of Life (QoL) assessment and treatment plan assessment, neither of which are known prior to consent. The post-inclusion criteria for the VITaL trial are:

1. Functional Assessment of Cancer Therapy - Lung (FACT-L) Trial Outcome Index (TOI) score of ≥5, the clinically meaningful difference
2. The standard treatment plan shows that at least 16% of volume of the lungs (minus the Gross Tumour Volume (GTV)) will receive more than 20 Gy. This criterion is based on the difference in pneumonitis risk between patients receiving below (~8%) and above (~34%) this threshold.

The QoL assessment is unlikely to eliminate any patients but is included for patients where no clinically meaningful difference will be possible. The treatment plan assessment may exclude 20% of otherwise eligible patients.

Exclusion Criteria:

1. Serious medical comorbidities that may contraindicate curative radiotherapy.
2. Inability to attend full course of radiotherapy or follow-up visits.
3. A current or former diagnosis of interstitial lung disease.
4. Prior history of lung cancer within 5 years.
5. Prior thoracic radiotherapy at any time.
6. Prior surgery for this cancer within a year.
7. Prior chemotherapy for this cancer.
8. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Patients receiving healthy lung sparing treatment (interventional arm) have better quality of life than patients receiving standard treatment (control arm). | 3 months
  Patients in the interventional healthy lung sparing arm will maintain their 3-month quality of life (measured via the Functional Assessment of Cancer Therapy - Lung (FACT-L) questionnaire) more than patients receiving standard care by a clinically meaningful difference.

SECONDARY OUTCOMES:
Interventional arm patients will have reduced treatment lung side-effects. | 2 years
  Toxicities will be collected at each patient visit.
Interventional arm patients will have better lung function, as determined by the difference between pre and post treatment Forced Expiratory Volume (FEV1) scores, as healthy lung is spared. | 2 years
  Lung function tests (FEV-1) will be acquired at routine time points within the trial, including pre and post treatment.
In the interventional arm, a higher proportion of patients will receive immunotherapy | 2 years
  Adjuvant therapy will be described for all patients as part of routine follow up.
In the interventional arm, a higher proportion of patients will complete immunotherapy | 2 years
  Adjuvant therapy will be described for all patients as part of routine follow up.
Cost effectiveness will be demonstrated as measured via a health economics assessment | 2 years
  To be determined

CONTACTS AND LOCATIONS:
Overall Officials: Paul Keall, PhD, Principal Investigator — University of Sydney
Locations (1):
- Liverpool Hospital, Liverpool, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
After study findings have been published, un-identifiable (non-coded, completely de-identified) data will be shared with researchers or at an external data repository for further scientific research.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be made available following the publication of the final results.
Access Criteria: Data will only be shared with repositories whose function has been reviewed and approved by an accredited Research Integrity/Ethics Committee/Board, under a Materials Transfer Agreement with the University of Sydney.